CLINICAL TRIAL: NCT02954133
Title: The Effect of OrthoPulse™ Photobiomodulation on Tooth Movement and Treatment Time When Used With Invisalign Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Biolux Research Holdings, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BX9
Record Dates: First submitted 2016-10-31; First posted 2016-11-03 (Estimated); Last update posted 2019-01-15 (Actual); Status verified 2019-01

CONDITIONS: Malocclusion
Keywords: Alignment phase; Photobiomodulation; Orthodontic treatment; Malocclusion; OrthoPulse™; Invisalign
MeSH Terms: conditions — Malocclusion | interventions — Orthodontic Appliances, Removable

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- I7: Control (Experimental): Subjects assigned to this group receive no OrthoPulse™ treatment, and switch Invisalign aligners every 7 days.
  Interventions: Device: Invisalign (7 day)
- OP7: OrthoPulse Treatment (Experimental): Subjects assigned to this group receive daily OrthoPulse™ treatments, and switch Invisalign aligners every 7 days.
  Interventions: Device: Invisalign (7 day); Device: OrthoPulse
- OP5: OrthoPulse Treatment (Experimental): Subjects assigned to this group receive daily OrthoPulse™ treatments, and switch Invisalign aligners every 5 days.
  Interventions: Device: Invisalign (5 day); Device: OrthoPulse
- OP3.5: OrthoPulse Treatment (Experimental): Subjects assigned to this group receive daily OrthoPulse™ treatments, and switch Invisalign aligners every 3.5 days.
  Interventions: Device: OrthoPulse; Device: Invisalign (3.5 day)

INTERVENTIONS:
Device: Invisalign (7 day) — Patients are are fitted with a ClinCheck plan by Align Technology by the qualified Principal Investigator (PI). Orthodontic treatment procedures carried out per the traditional practices of the PI and dental office. Aligners are switched every 7 days.
  Arms: I7: Control; OP7: OrthoPulse Treatment
Device: Invisalign (5 day) — Patients are are fitted with a ClinCheck plan by Align Technology by the qualified Principal Investigator (PI). Orthodontic treatment procedures carried out per the traditional practices of the PI and dental office. Aligners are switched every 5 days.
  Arms: OP5: OrthoPulse Treatment
Device: OrthoPulse — Daily 10 minute (5 minutes per arch) OrthoPulse treatments are administered at home.
  Arms: OP3.5: OrthoPulse Treatment; OP5: OrthoPulse Treatment; OP7: OrthoPulse Treatment
Device: Invisalign (3.5 day) — Patients are are fitted with a ClinCheck plan by Align Technology by the qualified Principal Investigator (PI). Orthodontic treatment procedures carried out per the traditional practices of the PI and dental office. Aligners are switched every 3.5 days.
  Arms: OP3.5: OrthoPulse Treatment

SUMMARY:
The aim of the study is to determine if, and to what degree photobiomodulation treatment with OrthoPulse has an effect on the rate of tooth movement during alignment for patients receiving Invisalign orthodontic aligner treatment.

ELIGIBILITY:
Inclusion Criteria:

* Invisalign "Full Treatment" product only
* Have a permanent dentition

  * 18 years-old
* Angle Class I or ½ cusp Class II molar and canine relationship
* Moderate to mild crowding in at least one arch

Exclusion Criteria:

* Subjects who do not fulfill all inclusion criteria requirements
* Craniofacial anomaly present
* Past or present signs and symptoms of periodontal disease
* A significant medical or medication history that would adversely affect the development or structure of the teeth and jaws and any subsequent tooth movement
* Previous orthodontic or orthopedic relapse within 1 year
* History of trauma, bruxism, or parafunction
* Skeletal jaw discrepancy
* Use of osteoporosis drugs
* Initial use of auxiliary mechanics such as elastics

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 167 (Actual)
Dates: Start 2016-07; Primary Completion 2019-04 (Estimated); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
Rate of tooth movement | From date of enrolment until the date of completion of the last Invisalign aligner, assessed every 4-6 weeks up to 2 years
  Tooth position will be measured at the end of aligners 6 (4-6 weeks), 12 (8-12 weeks), 18 (12-18 weeks), at the end first series of aligners at refinement, and at the end of treatment. Rates will be measured end of use of each individual Invisalign time point in order to determine whether the application of photobiomodulation increases the rate of tooth movement with Invisalign treatment.

SECONDARY OUTCOMES:
Length of treatment time | From date of enrolment until the date of completion of the last Invisalign aligner, assessed up to 2 years
  Treatment time will be calculated as the number of days from the first day until the last day the subject wears Invisalign aligners. To evaluate whether the application of photobiomodulation decreases the total treatment time with Invisalign treatment, the measured length of time will be compared against the expected treatment time.
Effect of photobiomodulation on external apical root resorption | From date of enrolment until the date of completion of the last Invisalign aligner, assessed up to 2 years
  Root lengths will be measured from panoramic radiographs to evaluate whether the application of photobiomodulation decreases the total amount of external apical root resorption over the course of the treatment,

CONTACTS AND LOCATIONS:
Overall Officials: Peter Brawn, DDS, Study Director — Biolux Research
Locations (4):
- United States (4):
  - Dickerson Orthodontics, Chandler, Arizona
  - Kottemann Orthodontics, Maple Grove, Minnesota
  - Chenin Orthodontics, Henderson, Nevada
  - Orthodontic Associates, Oklahoma City, Oklahoma

REFERENCES:
- [Background] Sun X, Zhu X, Xu C, Ye N, Zhu H. [Effects of low energy laser on tooth movement and remodeling of alveolar bone in rabbits]. Hua Xi Kou Qiang Yi Xue Za Zhi. 2001 Oct;19(5):290-3. Chinese. PMID 12539482
- [Background] Saito S, Shimizu N. Stimulatory effects of low-power laser irradiation on bone regeneration in midpalatal suture during expansion in the rat. Am J Orthod Dentofacial Orthop. 1997 May;111(5):525-32. doi: 10.1016/s0889-5406(97)70152-5. PMID 9155812
- [Background] Yamaguchi M, Hayashi M, Fujita S, Yoshida T, Utsunomiya T, Yamamoto H, Kasai K. Low-energy laser irradiation facilitates the velocity of tooth movement and the expressions of matrix metalloproteinase-9, cathepsin K, and alpha(v) beta(3) integrin in rats. Eur J Orthod. 2010 Apr;32(2):131-9. doi: 10.1093/ejo/cjp078. Epub 2010 Feb 16. PMID 20159792
- [Background] Nimeri G, Kau CH, Corona R, Shelly J. The effect of photobiomodulation on root resorption during orthodontic treatment. Clin Cosmet Investig Dent. 2014 Jan 15;6:1-8. doi: 10.2147/CCIDE.S49489. eCollection 2014. PMID 24470774
- [Background] Ekizer A, Uysal T, Guray E, Akkus D. Effect of LED-mediated-photobiomodulation therapy on orthodontic tooth movement and root resorption in rats. Lasers Med Sci. 2015 Feb;30(2):779-85. doi: 10.1007/s10103-013-1405-3. Epub 2013 Aug 29. PMID 23990217
- [Background] Ekizer A, Uysal T, Guray E, Yuksel Y. Light-emitting diode photobiomodulation: effect on bone formation in orthopedically expanded suture in rats--early bone changes. Lasers Med Sci. 2013 Sep;28(5):1263-70. doi: 10.1007/s10103-012-1214-0. Epub 2012 Nov 9. PMID 23139069
- [Background] El-Bialy T, Alhadlaq A, Felemban N, Yeung J, Ebrahim A, Hassan AH. The effect of light-emitting diode and laser on mandibular growth in rats. Angle Orthod. 2015 Mar;85(2):233-8. doi: 10.2319/030914-170.1. Epub 2014 Jul 14. PMID 25017014
- [Background] Uysal T, Ekizer A, Akcay H, Etoz O, Guray E. Resonance frequency analysis of orthodontic miniscrews subjected to light-emitting diode photobiomodulation therapy. Eur J Orthod. 2012 Feb;34(1):44-51. doi: 10.1093/ejo/cjq166. Epub 2010 Dec 27. PMID 21187526
- [Background] Kau CH, Kantarci A, Shaughnessy T, Vachiramon A, Santiwong P, de la Fuente A, Skrenes D, Ma D, Brawn P. Photobiomodulation accelerates orthodontic alignment in the early phase of treatment. Prog Orthod. 2013 Sep 19;14:30. doi: 10.1186/2196-1042-14-30. PMID 24326198
- [Background] Shaughnessy T, Kantarci A, Kau CH, Skrenes D, Skrenes S, Ma D. Intraoral photobiomodulation-induced orthodontic tooth alignment: a preliminary study. BMC Oral Health. 2016 Jan 13;16:3. doi: 10.1186/s12903-015-0159-7. PMID 26762247
- [Background] Doshi-Mehta G, Bhad-Patil WA. Efficacy of low-intensity laser therapy in reducing treatment time and orthodontic pain: a clinical investigation. Am J Orthod Dentofacial Orthop. 2012 Mar;141(3):289-297. doi: 10.1016/j.ajodo.2011.09.009. PMID 22381489
- [Background] Dias FJ, Issa JP, Vicentini FT, Fonseca MJ, Leao JC, Siessere S, Regalo SC, Iyomasa MM. Effects of low-level laser therapy on the oxidative metabolism and matrix proteins in the rat masseter muscle. Photomed Laser Surg. 2011 Oct;29(10):677-84. doi: 10.1089/pho.2010.2879. Epub 2011 Jul 11. PMID 21745137
- [Background] Silveira PC, Silva LA, Fraga DB, Freitas TP, Streck EL, Pinho R. Evaluation of mitochondrial respiratory chain activity in muscle healing by low-level laser therapy. J Photochem Photobiol B. 2009 May 4;95(2):89-92. doi: 10.1016/j.jphotobiol.2009.01.004. Epub 2009 Jan 21. PMID 19232497
- [Background] Cruz DR, Kohara EK, Ribeiro MS, Wetter NU. Effects of low-intensity laser therapy on the orthodontic movement velocity of human teeth: a preliminary study. Lasers Surg Med. 2004;35(2):117-20. doi: 10.1002/lsm.20076. PMID 15334614
- [Background] Youssef M, Ashkar S, Hamade E, Gutknecht N, Lampert F, Mir M. The effect of low-level laser therapy during orthodontic movement: a preliminary study. Lasers Med Sci. 2008 Jan;23(1):27-33. doi: 10.1007/s10103-007-0449-7. Epub 2007 Mar 15. PMID 17361391
- [Background] Sousa MV, Scanavini MA, Sannomiya EK, Velasco LG, Angelieri F. Influence of low-level laser on the speed of orthodontic movement. Photomed Laser Surg. 2011 Mar;29(3):191-6. doi: 10.1089/pho.2009.2652. Epub 2011 Jan 23. PMID 21254890
- [Background] Whelan HT, Smits RL Jr, Buchman EV, Whelan NT, Turner SG, Margolis DA, Cevenini V, Stinson H, Ignatius R, Martin T, Cwiklinski J, Philippi AF, Graf WR, Hodgson B, Gould L, Kane M, Chen G, Caviness J. Effect of NASA light-emitting diode irradiation on wound healing. J Clin Laser Med Surg. 2001 Dec;19(6):305-14. doi: 10.1089/104454701753342758. PMID 11776448
- [Background] Weber JB, Pinheiro AL, de Oliveira MG, Oliveira FA, Ramalho LM. Laser therapy improves healing of bone defects submitted to autologous bone graft. Photomed Laser Surg. 2006 Feb;24(1):38-44. doi: 10.1089/pho.2006.24.38. PMID 16503787
- [Background] Oron U, Ilic S, De Taboada L, Streeter J. Ga-As (808 nm) laser irradiation enhances ATP production in human neuronal cells in culture. Photomed Laser Surg. 2007 Jun;25(3):180-2. doi: 10.1089/pho.2007.2064. PMID 17603858